CLINICAL TRIAL: NCT07007455
Title: Effectiveness of Wrist Extensor Strength Training With Blood Flow Restriction on Lateral Elbow Tendinopathy
Acronym: BFR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, Shahnaz Hasan, PhD, Associate Professor, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUR
Record Dates: First submitted 2025-05-28; First posted 2025-06-05 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-01

CONDITIONS: Lateral Epicondylitis (Tennis Elbow); Elbow Pain; Lateral Elbow Tendinopathy; Extensor Carpi Radialis Brevis (ECRB)
Keywords: Wrist extensor strength training; lateral epicondylitis; Tennis elbow; elbow pain
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: This study will be a randomized controlled trial aimed at evaluating the effectiveness of wrist extensor strength training with blood flow restriction (BFR) in reducing pain, improving grip strength, and enhancing functional performance in individuals with lateral elbow tendinopathy.
Who Masked: Participant
Masking Description: Participants were randomly assigned to the experimental group (WEST-BFR) and the control group (WEST without BFR).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group: wrist extensor strength training with BFR. (Experimental): Experimental Group: Participants will undergo wrist extensor strength training with blood flow restriction (BFR).
  Interventions: Behavioral: wrist extensor strength training with BFR.
- Control Group: Wrist extensor strength training without BFR. (Active Comparator): Control Group: Participants will undergo the same wrist extensor strength training without blood flow restriction (BFR).
  Interventions: Behavioral: wrist extensor strength training without BFR.

INTERVENTIONS:
Behavioral: wrist extensor strength training with BFR. — Wrist extensor strength training without BFR.
  Other Names: Wrist extensor strength training without BFR.
  Arms: Experimental Group: wrist extensor strength training with BFR.
Behavioral: wrist extensor strength training without BFR. — wrist extensor strength training without BFR.
  Arms: Control Group: Wrist extensor strength training without BFR.

SUMMARY:
Repetitive and aggressive injuries to the elbow joint in sports often cause lateral elbow tendinitis (LET). In many clinical settings, therapists follow conventional methods according to their treatment protocols; however, complete rehabilitation is not always implemented. Without adequate care, elbow tendinitis can lead to chronic and recurring elbow injuries. Although many treatments are available, Blood flow restriction training (BFR) is a valuable option for exercise in cases where high-intensity training is too painful or contraindicated. In musculoskeletal disorders, it has been shown to induce hypoalgesia, and positive effects, such as improved muscle strength, growth, and tendon adaptations, have been demonstrated in healthy individuals.

DETAILED DESCRIPTION:
Lateral epicondylitis is a work-related musculoskeletal disorder and is defined as persistent symptomatic degeneration of the wrist extensor muscle tendon that connects to the lateral humeral epicondyle. It is characterized by pain on the lateral side of the elbow joint, limited range of motion, and weakness in the forearm muscles.

Management of lateral epicondylitis is aimed at reducing pain and discomfort, preserving ROM, and enhancing the strength and endurance of the affected limb by using numerous techniques, including electrophysical methods and physical activity.

Blood flow restriction training (BFRT) involves partially restricting arterial blood flow into muscles while occluding venous outflow during exercise. It was first introduced into the literature in 1987 by researchers who used tourniquet ischemia to induce fatigue in muscles, dating back to Dr. Yoshiaki Sato in Japan, where it was known as "kaatsu training," meaning "training with added pressure." Kaatsu training is now performed worldwide and is more commonly referred to as "BFR training," which is achieved using a pneumatic tourniquet system.

In addition to physical rehabilitation, BFRT is used for physical training and performance in healthy individuals. There has been extensive research into its value as a training tool, including elite- and amateur-level athletes, untrained young and older adults, and hypertensive individuals.

In addition to reducing arterial blood flow to working muscles, blood flow restriction obstructs venous return. When active muscles are exposed to BFR conditions, they are subjected to ischemia, which increases the metabolic stress on them. In addition to BFR, venous occlusion increases muscle cell swelling, activates intracellular anabolic pathways, and recruits fast-twitch fibers, which are thought to be involved in muscle adaptation.

There were different Factors affecting exercise adaptations with BFR, including pressure of occlusion (partial or complete), type of occlusion (continuous or intermittent), intensity of exercise, and volume of

Exercise with BFR:

BFR, along with low-load resistance training, cardio endurance training, and other activities that are generally recommended to improve muscular mass/strength, is also associated with these adaptations in muscles.

The randomized trial done by Karanasios et al to assess the effect of low-load resistance training with blood flow restriction (LLRT-BFR) versus LLRT with sham-BFR in patients with lateral elbow tendinopathy (LET) found that LLRT with blood flow restriction produced significantly better pain, strength, and function improvement in comparison to LLRT with sham-BFR for all primary outcomes(Karanasios et al., 2022).

Regarding the study of proximal and distal effects of BFR Training, a study by Bowman et al. on Lower extremity Low-load BFR training resulted in greater increases in muscle strength and limb circumference in healthy participants after completing a standardized 6-week course of BFR training. Muscle groups at the proximal and distal ends of the body were similarly strengthened after BFR training(Bowman et al., 2019).

This study aims to explore the effects of incorporating BFR into wrist extensor strength training for athletes with lateral epicondylitis. By evaluating its impact on strength, function, pain, range of motion (ROM), and overall quality of life, this research seeks to determine whether BFR can optimize rehabilitation outcomes and provide a more effective treatment strategy for LET.

ELIGIBILITY:
Inclusion Criteria:

1. Both Male and female, aged between 18 to 45 years old.
2. Subjects with a positive test of lateral epicondylitis, which will be determined based on physical therapy assessment procedures.
3. The presence of tenderness over the lateral epicondyle.positive Cozen's and Mill's tests.
4. Pain on grasping.
5. Pain on passive flexion of the wrist with elbow extension.
6. Pain with resisted wrist extension.
7. Show decreased muscle strength and functional ability.

Exclusion Criteria:

1. Patients with shoulder tendinopathy, cervical radiculopathy, and rheumatoid arthritis.
2. Presences of sensory and motor impairment of the upper extremities
3. History of cardiovascular disease
4. History of trauma and surgery on the elbow
5. Having a history of malignancy and peripheral vascular disorders.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 34 (Actual)
Dates: Start 2025-02-15 (Actual); Primary Completion 2025-05-15 (Actual); Study Completion 2025-05-25 (Actual)

PRIMARY OUTCOMES:
pressure pain thresholds (PPTs). | six weeks
  before and after intervention.
pain-free grip strength test | six weeks
  before and after intervention.

SECONDARY OUTCOMES:
Borg 6-20 scale | six weeks
  Participants will be asked to rate their effort after each set of exercises on a scale from 6 (no exertion) to 20 (maximal exertion).

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Health Rehabiltation Center, Al Majma'ah, Al Riyadh
  - Majmaah University, Al Majma'ah, Al-Riyadh

IPD SHARING:
Plan to Share IPD: Undecided
Not yet decided